CLINICAL TRIAL: NCT05173116
Title: Evaluation of API-VIGIE Monitoring System: Program to Reduce Emergency Visits for Severe Paroxysmal Alcoholism
Brief Title: Evaluation of the API-VIGIE Monitoring System: Program to Reduce Emergency Visits for Severe Paroxysmal Alcoholism
Acronym: EVAL-APIVIGIE
Status: Withdrawn | Type: Observational
Why Stopped: protocol not implemented for logistical reasons in the recruiting center, possible rescheduling.
Sponsor: Centre Hospitalier Arras (Other)
Collaborators: F2RSM Psy (Hauts-de-France Regional Federation for Research in Psychiatry and Mental Health) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-08
Record Dates: First submitted 2021-11-29; First posted 2021-12-29 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Intoxication;Alcohol;Acute; Emergencies
Keywords: Intoxication;Alcohol;Acute; Addiction, Alcohol; binge drinking; young adult
MeSH Terms: conditions — Alcoholic Intoxication; Emergencies; Alcoholism; Binge Drinking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prospective study: API-VIGIE program adult participant who agreed to participate in the study
  Interventions: Other: Medical Outcomes Study Short Form 36 (SF 36)
- retrospective study: Any stay for adults patients in the emergency room of the ARRAS hospital for API during the period covered (from 1 year before to 1 year after the installation of the APIVIGIE program) (main diagnosis or associated with an API (F10.0 according to the ICD-10 classification used by Department of Medical Information)
  Interventions: Other: observationnal study

INTERVENTIONS:
Other: Medical Outcomes Study Short Form 36 (SF 36) — completion of questionnaire quality of life SF 36 (inclusion, Month 3, Month 6).
  Groups: prospective study
Other: observationnal study — data collection
  Groups: retrospective study

SUMMARY:
The study was designed to evaluate the APIVIGIE program use at CH d'Arras. The objective of this program is to reduce repeated visits by the same patient to the emergency room for Alcoholism Severe Paroxysmal

DETAILED DESCRIPTION:
In France, between 10% and 30% of emergency room admissions are linked to problematic alcohol consumption. This considerable weight of alcohol-related problems in the current problematic of emergencies is largely unknown and can lead to blockages in emergencies.

For acute intoxication requiring emergency care, 80% of admissions concern people dependent on alcohol. Here again, this crucial clinical notion is largely ignored: when a patient in a state of intoxication arrives in the emergency room, this should not be considered as a banal and one-off event, it is necessary to put in place a care, if necessary, of addiction.

Supported by a call for projects from the Hauts-de-France Regional Health Agency, the Addictions Service of the Arras Hospital is setting up a monitoring system called APIVIGIE.

APIVIGIE program is offered to patients who present to the emergency room for a diagnosis of API after an evaluation by the liaison team of the addiction service. If the patient agrees to be part of the program, he will receive a resource card with the APIVIGIE phone number to contact if necessary.

The link will be maintained with the Addictology Care, Support and Prevention Center (CSAPA) for a period of 6 months, by telephone consultations, or by video-consultations or face-to-face consultations.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years or older;
* Participant at API-VIGIE program.

Exclusion Criteria:

* Patient's opposition to participating in the research;
* Persons under legal protection (under tutorship or curatorship);
* Person deprived of liberty;
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant at API-VIGIE program
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Number of visits to the Emergency Reception Service for Significant Paroxysmal Alcoholics | during 2 years
  1 year before implementation of the program and up to 1 year after implementation of the program

SECONDARY OUTCOMES:
weekly consumption of alcoholic beverages | Inclusion , Visit 2 (Month 3) and visit 3 (Month 6)
weekly consumption of other substances (cannabis, other substances) | Inclusion , Visit 2 (Month 3) and visit 3 (Month 6)
Quality of life score, measured by the Medical Outcomes Study Short Form 36 (SF-36) health scale score. | Inclusion , Visit 2 (Month 3) and visit 3 (Month 6)
  SF 36 giving a score from 0 to 100. More higher score, more better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique LEJEUNE, M.D, Principal Investigator — Centre Hospitalier Arras
Locations (1):
- Dominique LEJEUNE, Arras, France